CLINICAL TRIAL: NCT00003645
Title: A Phase III Randomized Prospective Trial of Adjuvant Hormonal Therapy in Surgically Treated Prostate Cancer Patients at High Risk for Recurrence
Brief Title: Randomized Trial of Adjuvant Hormonal Therapy in Surgically Treated Prostate Cancer Patients at High Risk for Recurrence
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per PI request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID97-077; P30CA016672 (NIH); MDA-ID-97077 (Other: UT MD Anderson Cancer Center); E-97077; NCI-T97-0069; CDR0000066733 (Registry Identifier: NCI PDQ); NCI-2009-00818 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 1999-11-01; First posted 2003-07-15 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Flutamide; Goserelin; Leuprolide; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Leuprolide + Flutamide (Experimental): Arm I: Patients receive leuprolide intramuscularly once every 3 months and oral flutamide three times daily for 1 year.
  Interventions: Drug: Flutamide; Drug: Leuprolide Acetate
- Arm II - No Treatment (No Intervention): Arm II: Patients receive no initial treatment.

INTERVENTIONS:
Drug: Flutamide — 10.8 mg intramuscularly once every 3 months for 12 months
  Other Names: Goserelin; Zoladex
  Arms: Arm I - Leuprolide + Flutamide
Drug: Leuprolide Acetate — 50 mg tablet orally daily for 12 months
  Other Names: Casodex; Bicalutamide
  Arms: Arm I - Leuprolide + Flutamide

SUMMARY:
RATIONALE: Testosterone can stimulate the growth of prostate cancer cells. Hormone therapy using leuprolide and flutamide may fight prostate cancer by reducing the production of testosterone. It is not yet known whether receiving leuprolide and flutamide is more effective than receiving no further therapy.

PURPOSE: Randomized phase III trial to determine the effectiveness of hormone therapy in treating patients who have stage I or stage II prostate cancer that is at high risk of recurrence and who have already undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of one year of adjuvant hormonal ablation on disease-free survival at 5 years in node-negative radical prostatectomy patients at high risk for progression.
* Determine the effect of this treatment on the incidence of androgen independent prostate cancer and on disease specific and overall survival.
* Determine the impact of one year of total androgen ablation on quality of life and serum testosterone levels.
* Assess differences in quality of life between wives of patients in the androgen ablation condition compared to wives of patients in the control condition.
* Obtain blood samples from patients at high risk for failure post-prostatectomy to evaluate serum markers of prognosis.

OUTLINE: This is a randomized study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive leuprolide intramuscularly once every 3 months and oral flutamide three times daily for 1 year.
* Arm II: Patients receive no initial treatment. Quality of life is assessed every 6 months for 5 years. Quality of life of wives/partners of patients is assessed every 6 months for two years.

Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

PROJECTED ACCRUAL: A total of 496 patients (248 per treatment arm) will be accrued for this study within 3.5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Organ confined prostate cancer (stage T1-T2c) subsequent to clinical staging
2. Radical prostatectomy and bilateral lymph node dissection performed
3. Pathologic assessment of surgical specimens by MDACC pathologist
4. High risk of clinical or biochemical failure post prostatectomy (must fulfill one of the following criteria): pathology; a) Gleason grade sum score greater than or equal to 8, b) Seminal vesicle involvement, c) Extraprostatic extension with positive surgical margins and Gleason greater than or equal to 7
5. Radical prostatectomy performed within 90 days of enrollment and serum PSA level < 0.1ng/ml
6. Written informed consent

Exclusion Criteria:

1. Any evidence of metastatic disease confirmed prior to enrollment
2. Inability to confirm pathologic risk factors or inadequate prostatectomy (see item 4.1.5).
3. Hormonal ablation for greater than 3 months or radiotherapy for prostate cancer
4. Failure to achieve prostate specific antigen level of less than 0.1ng/ml prior to enrollment in study
5. Elevation of liver function tests 2x normal
6. Contraindication to the use of LH-RH agonists or antiandrogens
7. Active secondary malignancy (other than squamous or basal cell skin cancer) within five years prior to enrollment in study
8. Any concomitant medical condition that would make it undesirable for the 7patient to participate in the trial or jeopardize compliance with the protocol

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1999-06-14 (Actual); Primary Completion 2017-03-20 (Actual); Study Completion 2017-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis A. Pettaway, MD, Study Chair — M.D. Anderson Cancer Center; Michael O. Koch, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study terminated early with low accrual with insufficient data for analysis.
Groups:
- Arm A: Goserelin + Bicalutamide (one year)
- Arm B: No initial treatment
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 30 | 34
Completed | 18 | 22
Not Completed | 12 | 12
Not completed — Death | 4 | 1
Not completed — Lost to Follow-up | 7 | 8
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 30 | 34 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 26 | 44
  >=65 years | 12 | 8 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 34 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 33 | 61
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 28 | 33 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 26 | 28 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 30 | 34 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease Free Survival at 5 Years
Description: To determine if one year of adjuvant hormonal ablation in node negative radical prostatectomy patients at high risk for progression will result in an improvement in disease-free survival at five years.
Time Frame: Beginning of the study up to 5 years
Population: The study terminated early without any participants reaching the 5 years on study analysis point.
Arm/Group | Arm I - Leuprolide + Flutamide | Arm II - No Treatment
Number analyzed (Participants) | 0 | 0

2. Other Pre Specified Outcome: Number of Wives of the Participants Having Better Than or Equal to a "Good" Quality of Life
Description: To measure the differences in quality of life between wives of participants in the androgen ablation condition compared to wives of patients in the control condition by using quality of life assessments. The following questionnaires were completed in the clinic setting and used to assess Health related (HRQoL): Medical Outcomes Study 36-Item Short Form (SF-36), University of California-Los Angeles Sexual Function Scale (UCLA-SFS), and Southwest Oncology Group Treatment-Specific Symptoms Scale (SWOG-TSSS). The SF-36 was analysed using a composite score for each of physical health and mental health. SF-36, UCLA-SFS, SWOGTSSS were combined to classify participants' quality of life.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 30 | 34
Participants | 19 | 24

3. Other Pre Specified Outcome: Quality of Life for Participants
Description: To determine the impact of one year of total androgen ablation on quality of life mentally, physically and sexual function. The following questionnaires were completed by patients in the clinic setting and used to assess HRQoL: Medical Outcomes Study 36-Item Short Form (SF-36) and University of California-Los Angeles Sexual Function Scale (UCLA-SFS). To score the SF-36, scales are standardized with a scoring algorithm or by the SF-36v2 scoring software to obtain a score ranging from 0 to 100. Higher scores indicate better quality of life.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm I - Leuprolide + Flutamide | Arm II - No Treatment
Number analyzed (Participants) | 21 | 22
score on a scale
  Mental | 55 [51 to 59] | 54 [52 to 57]
  Physical | 49 [44 to 54] | 49 [44 to 54]
  Sexual Function | 5 [0 to 8] | 28 [15 to 39]

4. Other Pre Specified Outcome: Markers of Prognosis
Description: To obtain blood/tissue samples from patients at high risk for failure post prostatectomy to evaluate markers of prognosis.
Time Frame: 1 year after treatment
Population: Due to poor study accrual there were not enough data collected to be analyzed to determine the markers of prognosis.
Arm/Group | Arm I - Leuprolide + Flutamide | Arm II - No Treatment
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 Year (duration of study treatment)
Description: AEs and SAEs were only assessed and documented for participants on treatment arm A
Arm/Group | Arm I - Leuprolide + Flutamide | Arm II - No Treatment
All-Cause Mortality (participants affected / at risk) | 4/30 | 1/34
Serious Adverse Events (participants affected / at risk) | 6/30 | 0/0
Other Adverse Events (participants affected / at risk) | 25/30 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Leuprolide + Flutamide (N=30) | Arm II - No Treatment (N=0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | NA
Infection (Infections and infestations) | 1 (1) | NA
DVT (Blood and lymphatic system disorders) | 1 (1) | NA
Chest Pain (Cardiac disorders) | 1 (1) | NA
Urinary Infection (Renal and urinary disorders) | 1 (1) | NA
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Leuprolide + Flutamide (N=30) | Arm II - No Treatment (N=0)
Fatigue (General disorders) | 17 (17) | NA
Hot Flashes (Vascular disorders) | 25 (25) | NA
Diarrhea (Gastrointestinal disorders) | 7 (7) | NA
Gynecomastia (Reproductive system and breast disorders) | 9 (9) | NA
Decreased Libido (Psychiatric disorders) | 8 (8) | NA
Skin Rash (Skin and subcutaneous tissue disorders) | 5 (5) | NA
Weight Gain (Investigations) | 4 (4) | NA
Insomnia (Psychiatric disorders) | 4 (4) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-07-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT00003645/Prot_SAP_000.pdf